CLINICAL TRIAL: NCT01451424
Title: A Phase 2, 3 Arm, Randomized, Double-Blind Study to Evaluate the Safety, PK and Efficacy of Proellex® Administered Vaginally in the Treatment of Premenopausal Women With Uterine Fibroids
Brief Title: Evaluation of Safety, Pharmacokinetics, and Efficacy of Proellex Administered Vaginally in Women With Uterine Fibroids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZPV-200
Record Dates: First submitted 2011-10-11; First posted 2011-10-13 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — telapristone acetate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Proellex 12 mg PK group (Experimental): Subjects receiving 12 mg Proellex administered vaginally, and completing a PK arm consisting of 1 x 24 hr PK of Proellex, 14 days of daily Proellex trough measurements, and 1 x 24 hr PK of Proellex after 14 days of daily dosing. 12 mg PK subjects will continue with the protocol as written after the first 2 week period and will be treated for a total of 16 weeks.
  Interventions: Drug: Proellex
- Proellex 12 mg per protocol (Experimental): Subjects receiving 12 mg Proellex daily, vaginally for 12 weeks
  Interventions: Drug: Proellex
- Proellex 6 mg per protocol (Experimental): Subjects receiving 6 mg Proellex daily, vaginally for 12 weeks
  Interventions: Drug: Proellex
- Proellex 3 mg per protocol (Experimental): Subjects will receive 3 mg Proellex daily, vaginally for 12 weeks.
  Interventions: Drug: Proellex
- 24 mg Proellex (Experimental): 24 mg vaginal Proellex daily for 16 weeks
  Interventions: Drug: Proellex

INTERVENTIONS:
Drug: Proellex — vaginal suppository, daily, for 12 weeks
  Other Names: Telapristone acetate

SUMMARY:
To determine the safety, pharmacokinetics and efficacy of 4 doses (3, 6, 12, 24 mg) of Proellex in premenopausal women with uterine fibroids confirmed by ultrasound. Drug will be administered vaginally.

DETAILED DESCRIPTION:
This study is a phase II, 5 arm study with a 12 week active dosing period. The study will be conducted in 2 stages. In the first stage, the first 6 women to be enrolled will be treated at the 12mg dose level, and in addition to the other required study assessments will be monitored with a 24-hour PK assessment on Day 14, and daily trough assessments for the first 14 days. If, at Visit 3, the Cmax or AUC of any subject treated at 12mg exceeds the mean observed for the highest safe oral dose administered in the ZP-204 study, all subjects enrolled at the 12mg level will be discontinued, no further patients will be treated at this dose level, and the 6mg vaginal dose will be assessed in a similar fashion. In the second stage, the remaining subjects will be randomized to a dose of 3, 6, 12 or 24 mg.

For all subjects there will be a 4-6 week placebo run-in period, to establish baseline parameters (bleeding and quality of life) followed by treatment at one of three single-blind Proellex doses (3, 6 or 12 mg daily, administered vaginally in capsule form.) The primary efficacy endpoint will be bleeding assessed using the Pictorial Blood Loss Assessment Chart (PBAC) after 12 or 16 weeks of treatment. The secondary endpoints will be changes in size of uterine fibroids assessed by MRI and improvement in quality of life assessed using the Uterine Fibroid Symptom and Health-Related Quality of Life questionnaire (UFSQOL0. Safety endpoints include significant adverse events, changes in physical examination results, and/or clinical laboratory results significantly outside of normal range. For subjects enrolled in Stage 2, PK will be assessed after the first and last doses and trough levels every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult females between 18 and 47 years of age with uterine fibroids confirmed by ultrasound.
* Normal transvaginal ultrasound (other than for presence of fibroids)
* History of menstrual events occurring in regular cycles
* Agreement not to attempt to become pregnant
* Agreement to limit alcohol consumption to no more than 2 drinks per week and to avoid alcohol consumption within 48 hours before each visit
* Ability to complete a daily subject diary
* Willing to discontinue hormonal contraceptives and consent to use of double barrier contraceptive techniques over the course of the study.
* Has a negative pregnancy test at the Screening and Baseline visits An exception for the pregnancy test requirement will be granted for subjects reporting surgical sterilization in medical history
* A Body Mass Index (BMI) between 18 and 39 inclusive
* Is available for all treatment and follow-up visits.

Exclusion Criteria:

* Subject is a post-menopausal woman, defined as either; six (6) months or more (immediately prior to screening visit) without a menstrual period, or prior hysterectomy and/or oophorectomy
* Subject is pregnant or lactating or is attempting or expecting to become pregnant during the 6 month study period
* Women with abnormally high liver enzymes or liver disease. (ALT or AST exceeding 1.5xULN AND total bilirubin exceeding 1.5xULN at screening and confirmed on repeat).
* Received an investigational drug in the 30 days prior to the screening for this study
* Women with a history of PCOS
* Concurrent use of any testosterone, progestin, androgen, estrogen, anabolic steroids, DHEA or hormonal products for at least 2 weeks prior to screening and during the study.
* Use of oral contraceptives in the preceding 2 weeks. Use of Depo-Provera® in the preceding 6 months.
* Has an IUD in place
* Women currently using narcotics
* Women currently taking spironolactone
* Infectious disease screen is positive for HIV or Hepatitis A, B or C
* Clinically significant abnormal findings on screening examination or any condition which in the opinion of the investigator would interfere with the participant's ability to comply with the study instructions or endanger the participant if she took part in the study

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D Wiehle, PhD, Study Director — Repros Therapeutics Inc.
Locations (2):
- United States (2):
  - Cetero Research, Miami Gardens, Florida
  - Advances in Health, Houston, Texas

REFERENCES:
- See also: Repros Therapeutics Inc corporate website — http://www.reprosrx.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Proellex 3 mg Per Protocol: Subjects will receive 3 mg Proellex daily, vaginally for 12 weeks.
  Proellex: vaginal suppository, daily, for 12 weeks
  All subjects completed the placebo run-in period and started active dosing.
- Proellex 6 mg Per Protocol: Subjects receiving 6 mg Proellex daily, vaginally for 12 weeks
  Proellex: vaginal suppository, daily, for 12 weeks
  All subjects completed the placebo run-in period and started active dosing.
- Proellex 12 mg Per Protocol: Subjects receiving 12 mg Proellex daily, vaginally for 12 or 16 weeks
  Proellex: vaginal suppository, daily, for 12 or 16 weeks
  The first 6 subjects dosed at 12 mg (arm 1, PK group) were dosed for 16 weeks, the second 6 (arm 3) were dosed for 12 weeks
  The first 6 subjects (arm 1) had no placebo run-in period. Arm 3 subjects all completed the placebo run-in period and started active dosing.
- 24 mg Proellex: 24 mg vaginal Proellex daily
  Proellex: vaginal suppository, daily, for 16 weeks
  All subjects completed the placebo run-in period and started active dosing.
Period: Overall Study
Arm/Group | Proellex 3 mg Per Protocol | Proellex 6 mg Per Protocol | Proellex 12 mg Per Protocol | 24 mg Proellex
Started | 9 | 9 | 12 | 10
Completed | 8 | 7 | 11 | 5
Not Completed | 1 | 2 | 1 | 5
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Proellex 12 mg Per Protocol: Subjects receiving 12 mg Proellex daily, vaginally for 12 or 16 weeks
  Proellex: vaginal suppository, daily, for 12 weeks Includes subjects from both arms 1 and 3 (PK group and non-PK groups)
- 24 mg Proellex: 24 mg vaginal Proellex daily
  Proellex: vaginal suppository, daily, for 16 weeks
- Total: Total of all reporting groups
Arm/Group | Proellex 3 mg Per Protocol | Proellex 6 mg Per Protocol | Proellex 12 mg Per Protocol | 24 mg Proellex | Total
Number analyzed (Participants) | 9 | 9 | 12 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (6.3) | 39.9 (6.9) | 39.8 (4.8) | 40.9 (5.2) | 39.8 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 12 | 10 | 40
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 12 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Vaginal Bleeding
Description: Change from baseline in vaginal bleeding assessed at the end of treatment (12 or 16 weeks) using a Pictorial Blood Loss Assessment Chart (PBAC), which measures volume (mL) of blood loss over a 28-day period
  Less blood loss represents an improvement.
Time Frame: 12 or 16 weeks
Population: MITT population
Measure: Median (Full Range); unit: mL
Groups:
- Proellex 12 mg Per Protocol: Subjects receiving 12 mg Proellex daily, vaginally for 12 or 16 weeks
  Proellex: vaginal suppository, daily, for 12 or 16 weeks
  The first 6 subjects dosed at 12 mg (arm 1) were dosed for 16 weeks, the second 6 (arm 3) were dosed for 12 weeks
Arm/Group | Proellex 3 mg Per Protocol | Proellex 6 mg Per Protocol | Proellex 12 mg Per Protocol | 24 mg Proellex
Number analyzed (Participants) | 8 | 7 | 10 | 4
mL | -83.5 [-102 to -4] | -36.0 [-124 to 266] | -63.5 [-242 to -14] | -39.5 [-201 to -17]

2. Secondary Outcome: Blood Levels of Proellex
Description: Determination of Cmax of Proellex at end of treatment
Time Frame: 12 or 16 weeks
Population: Subjects with end of treatment PK assessment
Measure: Mean (Standard Deviation); unit: ng/dL
Groups:
- Proellex 12 mg PK Group: Subjects receiving 12 mg Proellex administered vaginally, and completing a PK arm consisting of 1 x 24 hr PK of Proellex, 14 days of daily Proellex trough measurements, and 1 x 24 hr PK of Proellex after 14 days of daily dosing. 12 mg PK subjects will continue with the protocol as written after the first 2 week period.
  Proellex: vaginal suppository, daily, for 12 weeks
Arm/Group | Proellex 12 mg PK Group | Proellex 3 mg Per Protocol | Proellex 6 mg Per Protocol | Proellex 12 mg Per Protocol | 24 mg Proellex
Number analyzed (Participants) | 6 | 7 | 7 | 5 | 5
ng/dL | 11.1 (5.1) | 14.1 (6.6) | 11.6 (2.0) | 7.4 (5.3) | 10.2 (8.6)

3. Secondary Outcome: Uterine Fibroid Size
Description: Percent change in volume of confirmed uterine fibroids at end of treatment, assessed by MRI
Time Frame: 12 or 16 weeks
Population: MITT population
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Proellex 3 mg Per Protocol | Proellex 6 mg Per Protocol | Proellex 12 mg Per Protocol | 24 mg Proellex
Number analyzed (Participants) | 8 | 7 | 10 | 4
Percentage change | -9.9 [-50.7 to 35.8] | -13.4 [-28.1 to 21.3] | -21.9 [-42.8 to -9.6] | -3.5 [-61.5 to 11.5]

4. Secondary Outcome: Induction of Amenorrhea at End of Treatment
Description: Percentage of subjects with induced amenorrhea during last 28 days on drug
  Amenorrhea was deemed to be achieved if no daily bleeding score was greater than 1 during the last 28 calendar days of the dosing period. A score of 1 was to be indicated if spotting was observed which did not require a sanitary product. Subjects that terminated early were deemed not to have achieved amenorrhea.
Time Frame: End of treatment
Measure: Number; unit: Percentage of particpants
Arm/Group | Proellex 3 mg Per Protocol | Proellex 6 mg Per Protocol | Proellex 12 mg Per Protocol | 24 mg Proellex
Number analyzed (Participants) | 9 | 9 | 12 | 10
Percentage of particpants | 55.6 | 0 | 66.7 | 40.0

5. Secondary Outcome: Endometrial Thickness
Description: Percent change in median endometrial thickness from baseline to end of treatment assessed by ultrasound determination of uterine stripe.
Time Frame: 12 or 16 weeks
Population: Safety population, data based on subjects with both baseline and end of treatment assessments
Measure: Median (Full Range); unit: Percent change
Arm/Group | Proellex 3 mg Per Protocol | Proellex 6 mg Per Protocol | Proellex 12 mg Per Protocol | 24 mg Proellex
Number analyzed (Participants) | 9 | 6 | 12 | 4
Percent change | 60.8 [-38.1 to 144] | -25.8 [-83.8 to 746.2] | 39.3 [-52.7 to 243.8] | 32.3 [-64.3 to 116.7]

6. Secondary Outcome: Change in Quality of Life
Description: Percentage change from baseline in median quality of life using uterine fibroid symptom and quality of life questionnaire (UFSQOL)
Time Frame: 12 or 16 weeks
Population: MITT. Note: lower score is improvement
Measure: Median (Full Range); unit: Percent change
Arm/Group | Proellex 3 mg Per Protocol | Proellex 6 mg Per Protocol | Proellex 12 mg Per Protocol | 24 mg Proellex
Number analyzed (Participants) | 8 | 7 | 10 | 3
Percent change | -67.9 [-100.0 to 21.7] | -8.5 [-100.0 to 117.4] | -98.2 [-100.0 to -42.9] | -100.0 [-100.0 to -100.0]

ADVERSE EVENTS:
Description: The Proellex 12 mg Per Protocol Arm/Group includes both Stage 1 and Stage 2 participants, i.e. all subjects dosed at 12 mg
Groups:
- 24 mg Proellex: 24 mg vaginal Proellex daily
  Proellex: vaginal suppository, daily, for 12 weeks
Arm/Group | Proellex 3 mg Per Protocol | Proellex 6 mg Per Protocol | Proellex 12 mg Per Protocol | 24 mg Proellex
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/9 | 0/12 | 1/10
Other Adverse Events (participants affected / at risk) | 6/9 | 4/9 | 6/12 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proellex 3 mg Per Protocol (N=9) | Proellex 6 mg Per Protocol (N=9) | Proellex 12 mg Per Protocol (N=12) | 24 mg Proellex (N=10)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Subject treated at 6 mg, considered by PI to be probably related to treatment.
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Treated at 24 mg, considerd by PI to be unrelated to treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Proellex 3 mg Per Protocol (N=9) | Proellex 6 mg Per Protocol (N=9) | Proellex 12 mg Per Protocol (N=12) | 24 mg Proellex (N=10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Sleepiness (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0
Vaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal yeast infection (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Atypical squamous cells of undetermined significance (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Trichomonous vaginalis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tooth infection (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Rask (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1
Hot flashes (Vascular disorders) | 0 | 0 | 1 | 0
Tingling sensation both thighs (Nervous system disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1
Thyroid enlargement (Endocrine disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights